CLINICAL TRIAL: NCT03683849
Title: Dancing as Training Method for Fall Preventing in Patients Suffering From Osteoporosis
Brief Title: Dancing Against Fall Fractures in Osteoporosis Patients and Healthy Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Mikkel Jacobi Thomsen, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: MJT.PhD.2018-2021
Record Dates: First submitted 2018-09-18; First posted 2018-09-25 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Osteoporosis; Fall Injury
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dancing group (Experimental): Dance intervention group, inspired by the rhythm of Salsa. Training will be administered for an hour twice a week, for six months.
  Interventions: Other: Training
- Strength training group (Active Comparator): Strength training group. Training will be administered for an hour twice a week, for six months.
  Interventions: Other: Training
- Control (No Intervention): Control group

INTERVENTIONS:
Other: Training — One hour of training, twice a week, for six months.
  Arms: Dancing group; Strength training group

SUMMARY:
This study evaluates physiological measurements and their role in among falls in healthy elderly (65yr or older) or elderly suffering from osteoporosis. The study further seeks to evaluate if dancing can be used as training for preventing falls.

DETAILED DESCRIPTION:
This study seeks to examine the relationship between strength, postural control and bone mineral density on the risk of falling among elderly (65 yr or older). The study will carried out on osteoporosis patients and healthy, matched controls. The study further seeks to examine whether a dancing intervention may improve any of these parameters, resulting in a decreased risk of falling.

ELIGIBILITY:
Patient groups

Inclusion Criteria:

* Verified osteoporosis (T-score -2.5 to -3.5) from previous Dual-energy X-ray absorptiometry scanning (DXA)
* Receiving medical treatment for osteoporosis

Exclusion Criteria:

* Drug addiction defined as the use of cannabis, opioids or other drugs.
* Use of medical cannabis.
* Previous neurologic, musculoskeletal (besides osteoporosis) or mental illnesses
* Lack of ability to cooperate.
* Osteoporosis grade higher than moderate or severe (T-score < -3.5)

Healthy elderly groups

Inclusion Criteria:

• T-score higher than -2.5 from previous Dual-energy X-ray absorptiometry scanning (DXA)

Exclusion Criteria:

* Drug addiction defined as the use of cannabis, opioids or other drugs.
* Use of medical cannabis.
* Previous neurologic, musculoskeletal (besides osteoporosis) or mental illnesses
* Lack of ability to cooperate.
* Osteoporosis grade higher than mild, moderate or severe (T-score < -2.5)
* Receiving medical treatment for osteoporosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Falls | Changes from baseline at 6- and 18 months
  Number of falls

SECONDARY OUTCOMES:
Postural stability | Changes from baseline at 6- and 18 months
  Postural sway measured using a high resolution three-dimensional force platform
Pain intensity rating: McGill Pain Questionnaire | Changes from baseline at 6- and 18 months
  Pain on an 11-point numerical rating scale (0 = no pain, 10 = most intense pain imaginable), indicating pain areas on a body chart and filling out a McGill Pain Questionnaire
Physical Activity | Changes from baseline at 6- and 18 months
  Evaluation of physical activity using the Physical Activity Scale for Elderly (PASE) questionnaire
Fitness assessment | Changes from baseline at 6- and 18 months
  Evaluation of fitness using the Fullerton Functional Fitness Assessment. The test is a 6-item test. The score in each of the six tests is assessed separately and will not be used to provide a total score of the six tests.
Dynamical balance assessment | Changes from baseline at 6- and 18 months
  Evaluation of the dynamical balance using the Mini-Balance Evaluation Systems Test (Mini-BESTest), which is a 14-item test, scored on a 3-level ordinal scale. The scale ranges from 0-28, with a higher score representing better dynamical balance.
Bone mineral density | Changes from baseline at 18 months
  Bone mineral density (g/cm2) measured at spine (L1-L4) and hip, using a Hologic DXA scanner.
Gait variability | Changes from baseline at 6- and 18 months
  Kinematic analysis of gait, recorded using the Xsens system
Cognitive function | Changes from baseline at 6- and 18 months
  A n-back test is performed. Total number of substractions and number of mistakes made are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Jacobi Thomsen, PhD. stud., Principal Investigator — Aalborg University
Locations (1):
- SMI, Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomsen MJ, Liston M, Christensen MG, Vestergaard P, Hirata RP. Dancing Against falls iN Community-dwElling older adults (DANCE): a study protocol of a stratified, block-randomised trial. Inj Prev. 2022 Feb;28(1):93-101. doi: 10.1136/injuryprev-2021-044224. Epub 2021 Sep 20. PMID 34544808